CLINICAL TRIAL: NCT03580707
Title: Does BRV Have a Faster Onset Time and Greater Effect Than LEV in Epilepsy Patients?: A Prospective, Randomized, Crossover, Double-blind, Controlled Intravenous Study Using the PPR as a Pharmacodynamic Efficacy Endpoint
Brief Title: Does BRV Have Faster Onset Time & Greater Effect Than LEV in Epilepsy Pts Using PPR Pharmacodynamic Efficacy Endpoint
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Rosenfeld, William E., M.D. (Individual)
Collaborators: Comprehensive Epilepsy Care Center for Children & Adults (Other); Utrecht University (Other); PRA Health Sciences (Industry); UCB Biopharma S.P.R.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: SAIRB-18-0016
Record Dates: First submitted 2018-05-24; First posted 2018-07-09 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Photosensitive Epilepsy
MeSH Terms: conditions — Epilepsy, Reflex

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 (Active Comparator): Compare rapidity of CNS effects of levetiracetam (LEV) & brivaracetam (BRV) within same pt-(randomized, two-way crossover, dbl-blind in total 16 pts w/epilepsy. Pt 1: IV infusion over 15 min BRV will also be administered as 15-min.infusion. BRV vs LEV in randomized double blinded, crossover fashion.
  Interventions: Drug: BRV vs LEV in randomized double blinded, crossover fashion
- Part 2 (Active Comparator): Pt 2 Op I:Assuming statistically signify. diff. in rapidity of CNS action has been observed from an analysis of data set in Pt 1,will proceed w/ Pt 2Opt I. Levetiracetam (LEV) or brivaracetam (BRV administered in randomized, two-way crossover, dbl-blind design as IV infusion over 5 min. to another cohort of 8 pts w/photosensitive epilepsy OR Pt 2,Opt II: Assuming no statistically signif. diff. in rapidity of CNS action has been observed from an analysis of data set in Pt 1, will proceed w/Pt 2,Opt II. LEV or BRV will be administered, in randomized, two-way crossover, dbl-blind design as IV infusion over again 15 min. to another cohort of 8 pts w/ photosensitive epilepsy. LEV will be given as 500 mg dose & BRV as 25 mg dose. BRV vs LEV in randomized double blinded, crossover fashion.
  Interventions: Drug: BRV vs LEV in randomized double blinded, crossover fashion

INTERVENTIONS:
Drug: BRV vs LEV in randomized double blinded, crossover fashion — Single dose intravenous administration of BRV 100 mg over a 15 minutes period. On a subsequent occasion, (approximately 2 weeks later), the patient is crossed over to the other drug at a singular dose. On both occasions, intermittent photic stimulation is done 10 times in a two hour period. IPS is again conducted in the cross over portion as well. Coincident with IPS stimulation 10 blood samples will be drawn for BRV or LEV plasma concentration.
  Other Names: Intermit pho stim respect over 2 hours/each of 2 study days

SUMMARY:
The main purpose of this study is to see whether brivaracetam has a faster onset time and greater effect than levetiracetam in subjects with photosensitive seizures. Part 1 of the study will compare the effects of levetiracetam 1500 mg with the effects of brivaracetam 100 mg. Part 2, will compare the effects of levetiracetam 1500 mg with the effects of brivaracetam 100 mg or will compare the effects of levetiracetam 500mg with the effects of brivaracetam 25 mg.

DETAILED DESCRIPTION:
The proposed study in epilepsy patients with photosensitivity intends to extend the animal findings for the faster (and perhaps greater) pharmacodynamic effect of intravenous BRV versus LEV at equipotent doses. Doses and infusion times were chosen based on proven safety profiles of both drugs (UCB, data on file): maximal dose of 1500 mg LEV in 15 minutes (or in 5 minutes) and 100 mg for BRV (15 times more potency of BRV compared to LEV). The study proposes a comparison of the rapidity of the CNS effects of both LEV and BRV within the same patient (randomized, two-way crossover, double-blind in a total 16 patients with epilepsy 8 patients in Part 1 and 8 patients in Part 2) Study Part 1: an IV infusion over 15 minutes, appropriately diluted (per package insert for LEV); BRV will also be administered as a 15-minute infusion (anticipating similar language in the package insert for BRV);Study Part 2, Option I: Assuming a statistically significant difference in the rapidity of CNS action has been observed from an analysis of the data set in Study Part 1, will proceed with Study Part 2 Option I. LEV or BRV will be administered, in a randomized, two-way crossover, double-blind design as an IV infusion over 5 minutes, appropriately diluted, to another cohort of 8 patients with photosensitive epilepsy. (Potentially, a few of the same patients as under 'a' above could participate herein, if they are willing to repeat the study). OR Study Part 2, Option II: Assuming no statistically significant difference in the rapidity of CNS action has been observed from an analysis of the data set in Study Part 1, will proceed with Study Part 2, Option II. LEV or BRV will be administered, in a randomized, two-way crossover, double-blind design as an IV infusion over again 15 minutes, appropriately diluted, to another cohort of 8 patients with photosensitive epilepsy. (Potentially, a few of the same patients as under 'a' above could participate herein, if they are willing to repeat the study). However, LEV will be given as a 500 mg dose, and BRV as a 25 mg dose. Use of lower, nearly equipotent minimally effective doses of LEV and BRV will maximize ability to readily differentiate the electroencephalographic PPR effect between the two AEDs.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 65 years of age
* Male or female
* PPR at minimum at 60,50,40,30,25,20,18 or 16 Hz as upper threshold
* Drug naïve or at most with up to 4 AEDs, not being LEV or BRV

Exclusion Criteria:

* Current treatment with more than 4 AEDs
* LEV or BRV as current treatment or used in the previous month.
* History of severe side-effects or psychological side-effects with LEV or BRV use
* Being pregnant or insufficiently protected against pregnancy (see also ref 31) or lactating Female
* Serious internal medical disease (renal/hepatic/cardiovascular disease) as deemed by the on-site physician (WER)
* History of psychiatric disease that has been a reason for acute hospitalisation for their condition of depression, schizophrenia, mania, delirium or aggressive behaviour
* History of status epilepticus
* History of significant ethanol or illicit drug use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
"Comparison between Brivaracetam and Levetiracetam of the Time to Peak Effect (Abolition) and Time to >50% Diminution in Photo-Paroxysmal Response in Patients with Photosensitive Epilepsy" (1) | Six weeks
  Difference in time (minutes) required between drugs, BRV& LEV to abolish a PPR (photo-paroxysmal response on the pts encephalogram, EEG) after intermittent photic stimulation (IPS) tested in the same pt of 2 separate occasions. In Pt 1, 8 pts w/photosensitive epilepsy will be studied in double-blind, crossover fashion with 15-minute linear intravenous (i.v.) infusion of either 1500 mg LEV or BRV 100 mg as single dose. After 2 weeks, each pt will be tested in identical fashion w/opposite drug (crossover). Pt 2, Option 1, 8 pts w/photosensitive epilepsy will be studied in double-blind, crossover fashion. Same single mg doses of LEV and BRV will be used, but i.v. infusion time will be 5 minutes;primary outcome measure will be same.Part 2, Option 2, 8 pts w/photosensitive epilepsy will be studied in double-blind, crossover fashion. Single mg i.v. dose of 500 mg LEV or 25 mg BRV will be used, w/infusion time over 15 minutes;primary outcome measure will be the same.

SECONDARY OUTCOMES:
"Comparison between Brivaracetam and Levetiracetam of the Time to Peak Effect (Abolition) and Time to >50% Diminution in Photo-Paroxysmal Response in Patients with Photosensitive Epilepsy" (2) | Six weeks
  Difference in time (minutes) required between drugs,BRV & LEV to produce a >50% decrease in PPR (photo-paroxysmal response on pts encephalogram, EEG) after intermittent photic stimulation (IPS) tested in same pt of 2 separate occasions. Pt 1, 8 patients w/photosensitive epilepsy will be studied in double-blind, crossover fashion w/15-minute linear intravenous (i.v.) infusion of either 1500 mg LEV or BRV 100 mg as single dose. After 2 weeks, each pt will be tested in identical fashion w/opposite drug (crossover). In Pt 2, Option 1, 8 pts w/photosensitive epilepsy will be studied in double-blind, crossover fashion. Same single mg doses of LEV and BRV will be used, but i.v. infusion time will be 5 minutes; primary outcome measure will be the same. Pt 2, Option 2, 8 pts w/photosensitive epilepsy will be studied in double-blind, crossover fashion. Single mg i.v. dose of 500 mg LEV or 25 mg BRV will be used, with infusion time over 15 minutes; primary outcome measure will be same.

CONTACTS AND LOCATIONS:
Overall Officials: William E Rosenfeld, M.D., Principal Investigator — Comprehensive Epilepsy Care Center for Children & Adults
Locations (1):
- The Comprehensive Epilepsy Care Center For Children And Adults, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reed RC, Rosenfeld WE, Lippmann SM, Eijkemans RMJC, Kasteleijn-Nolst Trenite DGA. Rapidity of CNS Effect on Photoparoxysmal Response for Brivaracetam vs. Levetiracetam: A Randomized, Double-blind, Crossover Trial in Photosensitive Epilepsy Patients. CNS Drugs. 2020 Oct;34(10):1075-1086. doi: 10.1007/s40263-020-00761-1. PMID 32949370